CLINICAL TRIAL: NCT07272174
Title: Resistance Training and Cognitive Health in Perimenopause
Brief Title: Exercise in Perimenopause to Improve Cognitive Health
Acronym: EPIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H25-01552
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Perimenopause; Subjective Cognitive Complaints
Keywords: progressive resistance training, perimenopause
MeSH Terms: interventions — Pliability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Training (PRT) (Experimental): Each PRT session will be 1-hr in duration and consists of a warm-up (10 mins), PRT (45 mins), and cool-down (5 mins). 2x/week and group-based.
  Interventions: Behavioral: Progressive Resistance Training
- Balance, Flexibility, and Tone Exercises (BAT) (Active Comparator): Each BAT session will be 1-hr in duration. 2x/week and group-based.
  Interventions: Behavioral: Balance, Flexibility, and Tone Exercises

INTERVENTIONS:
Behavioral: Progressive Resistance Training — The sessions will occur in the Exercise Prescription Suite of the Centre for Aging SMART at VCH; this suite is a fully-equipped gym that includes treadmills, bikes, pneumatic resistance training equipment, and free weights. The training stimulus will initially be at 3 sets of 10-15 repetitions with proper form. At week 4, training intensity will progress from 60-82% of predicted 1 repetition maximum (RM) using the 8RM method. Every 4 weeks the 8RM test will be repeated.
  Other Names: PRT
  Arms: Progressive Resistance Training (PRT)
Behavioral: Balance, Flexibility, and Tone Exercises — Each BAT session will be 1-hr in duration and consist of Pilates mat exercises, Yoga-based poses and breathing, Kegel exercises, stretches, and relaxation techniques (e.g., visualization).
  Other Names: BAT
  Arms: Balance, Flexibility, and Tone Exercises (BAT)

SUMMARY:
Perimenopause is now considered a possible risk factor for dementia and may contribute to the fact that 2/3 of those living with Alzheimer's disease are females. Indeed, research studies show that middle-aged females demonstrate significant declines in their thinking abilities and detrimental changes in their brains as they go through perimenopause. Thus, perimenopausal females need strategies to bolster their brain health.

The World Health Organization strongly recommends physical activity interventions to reduce the risk of decline in thinking abilities. However, whether exercise can improve thinking abilities and brain health in perimenopausal females has not been examined. Our research aims to address this important knowledge gap in female brain health.

We will study the effects of a 6-month resistance exercise training (e.g., lifting free weights, exercise with weight machine) program on thinking abilities in 50 physically inactive perimenopausal females, aged 40 to 55 years, who are experiencing difficulties with their thinking abilities. In addition to measuring thinking abilities, we will determine if exercise benefits muscle health, heart health, sleep quality, psychological well-being, menopausal symptoms, and quality of life. We will also explore how resistance exercise training improves thinking abilities as such information can lead to new discoveries and therapies for brain health in females.

DETAILED DESCRIPTION:
1. PURPOSE:

   To determine if progressive resistance training (PRT) can improve cognitive outcomes compared to balance, flexibility, and tone (BAT) exercises in perimenopausal females aged 40-55 years with subjective cognitive complaints.
2. HYPOTHESIS:

   At the end of the intervention, PRT will result in an increase in words recalled during the RAVLT 20-minute delay vs no improve in BAT.
3. JUSTIFICATION:

   The menopause transition (MT) negatively impacts cognitive function and the brain. The majority of perimenopausal females experiences cognitive difficulties and have subjective cognitive complaints (SCCs). Verbal episodic memory and processing speed are most negatively impacted by the MT. Cognitive and brain changes during the MT can significantly impact career and financial wellbeing. The MT is thus a critical window to intervene for female brain health. Exercise can reduce dementia risk factors and promote cognitive health. No published randomized controlled trials have examined the effect of exercise on cognitive outcomes in perimenopausal females.
4. OBJECTIVE:

   To determine if 26 weeks of 2x/week progressive resistance training (PRT) can improve verbal episodic memory performance on the Rey Auditory Verbal Learning Test (RAVLT) compared with balance, flexibility, and tone exercises (BAT) for physically inactive perimenopausal females aged 40-55.
5. RESEARCH DESIGN:

A 26-week, assessor-blinded, two-arm, proof-of-concept trial with 50 physically inactive perimenopausal females, aged 40 to 55 years, with subjective cognitive complaints. Participants will be randomized 1:1 to PRT or BAT and measured at baseline, 13 weeks, and 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are biological females, as assigned at birth
* Are aged between 40 and 55 years
* Had at least 1 menstrual period in the last 10 months
* Are perimenopausal based on STRAW +10 Staging System, or answer "yes" to MQ6 questions of changes in periods, having hot flashes, or vaginal dryness, pain, or sexual concerns
* Have an intact uterus
* Have a Montreal Cognitive Assessment (MoCA) score >26/30, indicating normal cognition
* Have subjective cognitive complaints defined as responding "yes" to "Do you feel like your memory or thinking is becoming worse?"
* Completed high school education
* Read and speak English with acceptable visual and auditory acuity
* Are able to safely engage in moderate-intensity PRT as indicated by the PAR-Q+; and
* Are able to provide informed consent.

Exclusion Criteria:

* Are engaged in regular PRT (i.e., 2x/week) in the prior three months
* Are diagnosed with cognitive impairment or dementia of any type
* Are at high risk for cardiac complications during exercise
* Have clinically important peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility
* Are taking medications that negatively affect cognitive function, such as anticholinergics, major tranquilizers, and anticonvulsants
* Have a BMI <15 or anorexia nervosa; g) had surgical menopause
* Had endometrial ablation that resulted in the loss of menstruation
* Have polycystic ovarian syndrome
* Currently undergoing chemo
* Had premature ovarian failure; or
* Are already enrolled in a drug or exercise trial

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test (RAVLT) | Baseline, 13 weeks, 26 weeks
  The RAVLT is a valid, reliable, and widely-used instrument of verbal episodic memory and learning, with normative values.

SECONDARY OUTCOMES:
NIH TB Cognitive Battery - Flanker Test | Baseline, 13 weeks, 26 weeks
  A measure of executive functions
NIH TB Cognitive Battery - Dimensional Change Card Sort Test | Baseline, 13 weeks, 26 weeks
  A measure of executive functions
NIH TB Cognitive Battery - Picture Sequence Memory Test | Baseline, 13 weeks, 26 weeks
  A measure of visual episodic memory
NIH TB Cognitive Battery - List Sorting Test | Baseline, 13 weeks, 26 weeks
  A measure of working memory
NIH TB Cognitive Battery - Pattern Comparison Processing Speed Test | Baseline, 13 weeks, 26 weeks
  A measure of processing speed
Everyday Memory Questionnaire | Baseline, 13 weeks, 26 weeks
  A subjective measure of memory failure in everyday life
Muscle strength of quads | Baseline, 13 weeks, 26 weeks
  Muscle strength measure by isokinetic dynamometer
Peripheral QCT of the tibia | Baseline, 13 weeks, 26 weeks
  A measure of bone and muscle health
Blood pressure | Baseline, 13 weeks, 26 weeks
  Blood pressure - systolic and diastolic
Lipid panel | Baseline, 26 weeks
  Lipid levels
Hemoglobin A1-C | Baseline, 26 weeks
  Average blood sugar levels
C-reactive protein | Baseline, 26 weeks
  Measure of inflammation
Health resource utilization | Baseline, 13 weeks, 26 weeks
  Cost of health resource used
Carotid-femoral pulse wave velocity | Baseline, 13 weeks, 26 weeks
  Arterial stiffness
Pittsburgh Sleep Quality Index | Baseline, 13 weeks, 26 weeks
  Subjective sleep quality
Sensewear Band | Baseline, 13 weeks, 26 weeks
  Using actigraphy data, quantify sleep quality (e.g., duration, efficiency, fragmentation).
Sensewear Band | Baseline, 13 weeks, 26 weeks
  Using actigraphy data, quantify physical activity (e.g., intensity and minutes)
Sensewear Band | Baseline, 13 weeks, 26 weeks
  Using actigraphy data, quantify sedentary behaviour (minutes)
Fatigue Severity Scale | Baseline, 13 weeks, 26 weeks
  Subjective fatigue
PHQ-9 | Baseline, 13 weeks, 26 weeks
  Depression severity
GAD-7 | Baseline, 13 weeks, 26 weeks
  Generalized anxiety disorder
Menopause Rating Scale | Baseline, 13 weeks, 26 weeks
  Menopause symptoms
EuroQol-5 Domain-5 Level | Baseline, 13 weeks, 26 weeks
  Quality of life
International Physical Activity Questionnaire | Every 30 days over 26 weeks
  Physical activity
DEXA | Baseline, 13 weeks, 26 weeks
  Lean mass
DEXA | Baseline, 13 weeks, 26 weeks
  Body fat
DEXA | Baseline, 13 weeks, 26 weeks
  Appendicular Skeletal Muscle Mass Index (ASMI); a measure of sarcopenia
Mediterranean-DASH Diet Intervention for Neurodegenerative Delay (MIND) Diet score | Baseline, 13 weeks, 26 weeks
  Diet
Processing Speed by smartphone | Baseline, 13 weeks, 26 weeks
  Processing Speed
Memory by smartphone | Baseline, 13 weeks, 26 weeks
  Memory
Productivity Questionnaire | Baseline, 13 weeks, 26 weeks
  Measure of work productivity
Brain-Derived Neurotrophic Factor | Baseline, 26 weeks
  Neurotrophic Factor
IGF-1 | Baseline, 26 weeks
  Neurotrophic Factor

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No